CLINICAL TRIAL: NCT01092728
Title: A Phase II Study of Biological Response to Dasatinib Treatment in Patients With Acral Lentiginous, Mucosal, or Chronic Sun-damaged Melanoma
Brief Title: Treatment With Dasatinib in Patients With Acral Lentiginous, Mucosal, or Chronic Sun-damaged Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0447; NCI-2011-00468 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-03-23; First posted 2010-03-25 (Estimated); Results first posted 2016-09-05 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-07

CONDITIONS: Melanoma
Keywords: Acral lentiginous melanoma; Mucosal melanoma; Chronic sun-damaged melanoma; Surgically removed tumor; biopsied; Sprycel; Dasatinib
MeSH Terms: conditions — Melanoma | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1: Completely Resectable (Active Comparator): Dasatinib 100 mg daily for 7 days and then surgical resection on Day 8. Afterwards, Dasatinib 100 mg daily will be administered for a total of 12 months/12 cycles (1 cycle = 4 weeks of treatment).
  Interventions: Drug: Dasatinib; Procedure: Surgical Resection
- Group 2: Unresectable (Active Comparator): 100 mg Dasatinib daily continued up to 12 months/12 cycles (1 cycle = 4 weeks of treatment).
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib — 100 mg daily.
  Other Names: BMS-354825; Sprycel
Procedure: Surgical Resection — Complete surgical resection of tumor(s).
  Arms: Group 1: Completely Resectable

SUMMARY:
The goal of this clinical research study is to compare how the drug Sprycel (dasatinib) can help to control the tumor in Patients With Acral Lentiginous, Mucosal, or Chronic Sun-damaged Melanoma. The safety of this drug will also be studied.

Objectives:

Primary Objectives:

1. To compare the biological response of tumors With and Without Resectable Tumors from patients with acral, or mucosal melanomas after treatment with dasatinib.

Secondary Objectives:

1. To assess the safety and tolerability of dasatinib in this patient population

   Completely Resectable Acral, Chronic Sun-damaged (CSD), and Mucosal Melanoma:
2. To assess the median time to recurrence and overall survival of patients with completely resectable acral, CSD, and mucosal melanoma treated with dasatinib
3. To assess whether FDG-avidity and KIT phosphorylation responses after treatment with dasatinib predicts prolonged time to recurrence and/or overall survival in patients with completely resectable acral, CSD, and mucosal melanomas

   Not Completely Resectable Acral, CSD, and Mucosal Melanoma:
4. To assess the response rate, progression free survival, and overall survival of patients with acral, CSD, and mucosal melanoma treated with dasatinib
5. To assess whether FDG-avidity and KIT phosphorylation responses after treatment with dasatinib predicts response rate, progression free survival, and/or overall survival in patients with acral, CSD, and mucosal melanomas

DETAILED DESCRIPTION:
The Study Drug:

Dasatinib is designed to change the function of genes. By changing the function of these genes, it may prevent cancer from growing and spreading.

Study Groups:

If you are found to be eligible to take part in this study, you will be placed into one of two groups depending on if the disease can be removed by surgery on or not. Group 1 will be patients who have melanoma that can be removed by surgery. Group 2 will be patients who have melanoma that cannot be completely removed by surgery.

Study Drug Administration:

For this study, every 4 weeks is a study "cycle."

Dasatinib pills will be taken by mouth with a full glass (8 ounces) of water with or without a meal. The pills should not be crushed or cut, they should be swallowed whole.

If you are in Group 1, you will take 2 dasatinib pills 1 time every day, for 7 days before your already-scheduled surgery. About 6 weeks after surgery (depending on how long it takes you to recover) you will begin taking 2 dasatinib pills 1 time every day for up to 13 cycles as long as you tolerate it and the disease does not come back.

If you are in Group 2, you will take 2 dasatinib pills 1 time every day, for 7 days before your already-scheduled biopsy on Day 8 (+/1 business day) of Cycle 1. Within 5 days after the biopsy, you will begin taking 2 dasatinib pills 1 time every day for up to 13 cycles, as long as you tolerate it and the disease does not come back.

Both groups will be given a pill chart to fill out at home to record when you take the study drug, and how many pills you take each time. You will need to bring the pill chart to every study visit for the study doctor to review. You will also need to bring the pill bottles to each study visit.

Group 1 Study Visits:

After the screening tests have been complete, and before you start taking the study drug, the following procedures will be performed:

* Your weight and vital signs will be measured.
* You will be asked about any drugs you may be taking.
* Your performance status will be recorded.

After 7 days of taking the study drug, and before surgery, the following procedures will be performed:

* You will have a physical exam, including a measurement of your weight and vital signs.
* Blood (about 1 tablespoon) will be drawn for routine tests.
* Your performance status will be recorded.
* You will be asked about any other drugs you may be taking.
* You will have an ECG to check your heart function.
* You will have a PET scan to check the status of the disease.

About 6 weeks after surgery, when you begin taking the study drug on Cycle 1, the following tests and procedures will be performed on Day 1 of each cycle:

* Blood (about 1 tablespoon) will be drawn for routine tests.
* You will have a physical exam, including a measurement of your weight and vital signs.
* Your performance status will be recorded.
* You will be asked about any other drugs you may be taking, and any side effects you may be experiencing.

On Day 15 of Cycle 1 only, the following tests and procedures will be performed:

* Blood (about 1 tablespoon) will be drawn for routine tests.
* You will have a physical exam, including a measurement of your weight and vital signs.
* Your performance status will be recorded.
* You will be asked about any other drugs you may be taking, and any side effects you may be experiencing.

Every 12 weeks while you are receiving treatment, the following tests and procedures will be performed:

* An ECG will be performed to check your heart function.
* You will have a CT scan or MRI scan of the chest, abdomen, and pelvis to check the status of the disease.

Group 2 Study Visits:

After the screening tests have been complete, and before you start taking the study drug, the following procedures will be performed:

* You will have a measurement of your vital signs including your weight.
* You will be asked about any drugs you may be taking.
* Your performance status will be recorded.

After 7 days of taking the study drug, and before the biopsy, the following procedures will be performed:

* You will have a physical exam, including a measurement of your weight and vital signs.
* Blood (about 1 tablespoon) will be drawn for routine tests.
* Your performance status will be recorded.
* You will be asked about any other drugs you may be taking.
* You will have an ECG to check your heart function.
* You will have a PET scan to check the status of the disease.

About 5 days after the biopsy, you will begin taking the study drug again for 3 more weeks to complete Cycle 1. On Day 15 of Cycle 1 only, the following tests and procedures will be performed:

* Blood (about 1 tablespoon) will be drawn for routine tests.
* You will have a physical exam including a measurement of your weight and vital signs.
* Your performance status will be recorded.
* You will be asked about any other drugs you may be taking, and any side effects you may be experiencing.

The following tests and procedures will be performed on Day 1 of each cycle starting with Cycle 2:

* Blood (about 1 tablespoon) will be drawn for routine tests.
* You will have a physical exam, including a measurement of your weight and vital signs.
* Your performance status will be recorded.
* You will be asked about any other drugs you may be taking, and any side effects you may be experiencing.

Every 12 weeks while you are receiving treatment, the following tests and procedures will be performed:

* An ECG will be performed to check your heart function.
* You will have a CT scan or MRI scan of the chest, abdomen, and pelvis to check on the status of the disease.

Length of Study:

You will continue to take the study drug for up to 13 cycles. You will be taken off study early if you experience intolerable side effects, the disease returns (Group 1 only), the disease gets worse (Group 2 only), or if the study doctor thinks it is in your best interest.

If you are in Group 2, and you are benefiting from the treatment, you may be allowed to continue to receive treatment with the study drug after you have completed the 12 study cycles. The study doctor will discuss this option with you in more detail.

End-of-Study Visit:

Within 30 days after the last dose of study drug, you will have an end-of-study visit, at which the following tests and procedures will be performed:

* Blood (about 1 tablespoon) will be drawn for routine tests.
* An ECG will be performed to check your heart function.
* You will have a CT scan or MRI scan of your chest, abdomen, and pelvis performed to check the status of the disease.
* You will have a physical exam, including a measurement of your weight and vital signs.
* Your performance status will be recorded.
* You will be asked about any other drugs you may be taking, and any side effects you may be experiencing.

Follow-Up Visits:

After your participation on this study is complete, you will have follow-up visit every 3 months and you will be asked about your health status. If you do not come to the hospital for a regularly scheduled clinic visit, you will receive a follow-up phone call. The phone call should last about 15 minutes each time.

This is an investigational study. Dasatinib is FDA approved and commercially available for the treatment of certain types of leukemia. The use of dasatinib to treat acral lentiginous melanoma, mucosal melanoma, or chronic sun-damaged melanoma is investigational.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have primary, recurrent or metastatic melanoma with one of the following pathology or characteristics: i) acral lentiginous melanoma ii) mucosal melanoma iii) any known KIT mutation.
2. (Continued 1) If 20 patients without tumors harboring exon 11 or 13 KIT mutation are enrolled and treated before the completion of the patient accrual of 30, only those with tumors harboring exon 11 or 13 KIT mutation will be enrolled. Likewise, if 10 patients with tumors harboring exon 11 or 13 KIT mutation are enrolled and treated before the completion of the patient accrual of 30, only those without tumors harboring exon 11 or 13 KIT mutation will then be enrolled.
3. Patients must have measurable disease by 18-Fluoro-deoxyglucose positron emission tomography (FDG-PET) (with or without computed tomography (CT)) defined as having a maximum standardized uptake value (SUVmax) of 3 and SUVmax ofat least 2 fold greater than background.
4. Patients scheduled for FDG-PET should have uptake of the tracer in at least one lesion (tumor-to-muscle ratio >2) in the baseline PET/CT scan in order to be eligible for the follow-up FDG PET scans.
5. Patient must have surgically resectable melanoma lesion(s) or biopsiable lesion(s) which are amenable to 2 separate biopsy procedures by a core needle or excision.
6. Age >/= 18 years.
7. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
8. Adequate Organ Function: a. Total bilirubin < 2.0 times the institutional Upper Limit of Normal (ULN), b.Hepatic enzymes (aspartate transaminase, alanine transaminase (AST, ALT) ) </= 2.5 times the institutional ULN, c. Serum Creatinine < 1.5 time the institutional ULN, d.Neutrophil count >/= 1500; Platelets >/= 75,000;
9. Ability to take oral medication (dasatinib must be swallowed whole)
10. Concomitant Medications: a. Patient agrees to discontinue St. Johns Wort while receiving dasatinib therapy (discontinue St. Johns Wort at least 5 days before starting dasatinib), b.Patient agrees that IV bisphosphonates will be withheld for the first 8 weeks of dasatinib therapy due to risk of hypocalcemia.
11. Women of childbearing potential (WOCBP) must have: a) A negative serum or urine pregnancy test (sensitivity 25 IU human chorionic gonadotropin (HCG/L) within 72 hours prior to the start of study drug administration b) Persons of reproductive potential must agree to use and utilize an adequate method of contraception throughout treatment and for at least 4 weeks after study drug is stopped. Prior to study enrollment, women of childbearing potential must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy.
12. Signed written informed consent including a Health Insurance Portability and Accountability Act (HIPAA) form according to institutional guidelines

Exclusion Criteria:

1. No other malignancy which required radiotherapy or systemic treatment within the past 5 years.
2. Concurrent medical condition which may increase the risk of toxicity, including: a. Pleural or pericardial effusion of any grade.
3. Cardiac Symptoms; any of the following should be considered for exclusion: a. Uncontrolled angina, congestive heart failure or MI within (6 months), b. Diagnosed congenital long QT syndrome, c. Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes), d. Prolonged corrected QT interval (QTc) interval on pre-entry electrocardiogram (> 480 msec) [or > 500 msec for patients with a bundle branch block]), e. Subjects with hypokalemia or hypomagnesemia if it cannot be corrected prior to dasatinib administration.
4. History of significant bleeding disorder unrelated to cancer, including: a. Diagnosed congenital bleeding disorders (e.g., von Willebrand's disease), b. Diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies), c. Ongoing or recent (</= 3 months) significant gastrointestinal bleeding.
5. Concomitant Medications, any of the following should be considered for exclusion: a. Category I drugs that are generally accepted to have a risk of causing Torsades de Pointes including: (Patients must discontinue drug 7 days prior to starting dasatinib), I. quinidine, procainamide, disopyramide, II. amiodarone, sotalol, ibutilide, dofetilide, III. erythromycin, clarithromycin, IV. chlorpromazine, haloperidol, mesoridazine, thioridazine, pimozide V. cisapride, bepridil, droperidol, methadone, arsenic, chloroquine, domperidone, halofantrine, levomethadyl, pentamidine, sparfloxacin, lidoflazine.
6. Women who: a. are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for at least 4 weeks after cessation of study drug, or, b. have a positive pregnancy test at baseline, or, c. are pregnant or breastfeeding,
7. Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious) illness
8. No active, untreated brain metastases. Patients with known brain metastases will be included if the brain metastases have been treated and stable for at least 3 months without the use of steroid
9. HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with dasatinib. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
10. Patients with melanoma harboring BRAF mutation. If BRAF mutation is not known at the time of screening, patients will still be eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-03; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin B. Kim, MD, BA, Study Chair — UT MD Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: March 2011 to September 2013. All recruitment was done at The University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: A total of 19 participants were enrolled, out of which 18 participants were included in the analysis and 1 participant was a screen failure.
Groups:
- Dasatinib + Completely Resectable: Participants will receive Dasatinib 100 mg daily for 7 days. Surgical Tumor Resection on Day 8. Afterwards, Dasatinib 100 mg daily will be administered for a total of 12 months/12 cycles (1 cycle = 4 weeks of treatment).
- Dasatinib + Unresectable: Dasatinib 100 mg daily will be administered for a total of 12 months/12 cycles (1 cycle = 4 weeks of treatment).
Period: Overall Study
Arm/Group | Dasatinib + Completely Resectable | Dasatinib + Unresectable
Started | 4 | 14
Completed | 0 | 0
Not Completed | 4 | 14
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Disease Progression | 1 | 13
Not completed — Prohibited Concomitant Medications | 1 | 0

BASELINE CHARACTERISTICS:
Population: One participant was screen-failed prior to study group entry.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dasatinib + Completely Resectable | Dasatinib + Unresectable | Total
Number analyzed (Participants) | 4 | 14 | 18
Age, Continuous [Median (Full Range); unit: years] | 76 [74 to 81] | 66 [43 to 79] | 71 [43 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 10 | 12
  Male | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 4 | 14 | 18

OUTCOME MEASURES:

1. Primary Outcome: Biologic Response Evaluation of Tumors With and Without Resectable Tumors
Description: Biologic response defined as either (complete or partial) metabolic tumor response after 7 days dasatinib treatment by positron emission tomography (PET) scan, >/= 25% decrease in Fluorodeoxyglucose (FDG) activity on PET without >15% increase in tumoral Ki-67 expression or >/=25% decrease in tumoral Ki-67 expression without >15% increase in FDG activity on PET scan. Complete Metabolic Response (CMR): FDG-avidity all lesions reduced to background FDG-avidity level. Partial Metabolic Response (PMR): >/=25% decrease in FDG-avidity as represented by change in mean Standardized Uptake Values (SUV) max. SUVmax measured by drawing region of interest slightly outside each lesion corresponding to those on CT image & adjusted for body weight. Measureable disease by PET scan defined as lesions that can be determined to have FDG-avidity of SUVmax of 3 and 2 x background.
  PR or CR confirmatory disease assessment performed >4 weeks (28 days) after criteria for response first met.
Time Frame: Assessment at 7 Days with confirmatory disease assessment performed no less than 4 weeks (28 days) afterwards
Population: Of 4 participants in first arm, none were evaluable for response (1 inevaluable, 2 withdrawals, 1 disease progression); and of the second arm, one was inevaluable (withdrawal).
Measure: Number; unit: participants
Arm/Group | Dasatinib + Completely Resectable | Dasatinib + Unresectable
Number analyzed (Participants) | 0 | 13
participants
  Complete Metabolic Response |  | 0
  Partial Metabolic Response |  | 1

2. Secondary Outcome: Progression-Free Survival
Description: Progression-Free Survival (PFS) is defined as the duration of time from start of treatment to date of first evidence of progression or the date of last follow-up for patients who do not progress.
Time Frame: Evaluated every 2 cycles (8 weeks) until disease progression or last follow-up, up to two years
Population: None of the participants in the Resectable arm were evaluable, and one participant in the second Unresectable arm was inevaluable due to early departure from study.
Measure: Median (Full Range); unit: Weeks
Arm/Group | Dasatinib + Completely Resectable | Dasatinib + Unresectable
Number analyzed (Participants) | 0 | 13
Weeks |  | 8.00 [0.86 to 89.57]

ADVERSE EVENTS:
Time Frame: Adverse events (AE)s and Serious Adverse Events (SAE)s were collected throughout the study from informed consent until 30 days after study treatment was discontinued. Overall AE collection period: March 11, 2011 to September 09, 2013.
Arm/Group | Dasatinib + Completely Resectable | Dasatinib + Unresectable
Serious Adverse Events (participants affected / at risk) | 0/4 | 4/14
Other Adverse Events (participants affected / at risk) | 4/4 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dasatinib + Completely Resectable (N=4) | Dasatinib + Unresectable (N=14)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dehydration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dasatinib + Completely Resectable (N=4) | Dasatinib + Unresectable (N=14)
Platelet Count Decreased (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Vaginal Hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Hemoglobin Decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Edema Limbs (Blood and lymphatic system disorders) | 0 (0) | 7 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 8 (11)
Blood Glucose Increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 7 (8)
Headache (General disorders) | 1 (1) | 9 (10)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 8 (10)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Neutrophil Count Decreased (Blood and lymphatic system disorders) | 0 (0) | 1 (4)
Insomnia (General disorders) | 0 (0) | 2 (2)
Serum Potassium Decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (6)
Anorexia (Gastrointestinal disorders) | 0 (0) | 6 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (7)
Weight Gain (General disorders) | 1 (1) | 3 (3)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 7 (8)
Vomiting (Gastrointestinal disorders) | 1 (1) | 5 (5)
Pain (General disorders) | 2 (2) | 3 (3)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 5 (6)
Rash Desquamating (Skin and subcutaneous tissue disorders) | 0 (0) | 6 (7)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constitutional Symptoms (General disorders) | 1 (1) | 2 (2)
Chest Pain (General disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 2 (2)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Confusion (Nervous system disorders) | 0 (0) | 1 (1)
Localized Edema (General disorders) | 0 (0) | 1 (1)
Hemorrhage/Bleeding (Vascular disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vaginal Infection (Infections and infestations) | 0 (0) | 1 (1)
Fatigue (General disorders) | 4 (4) | 12 (18)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes